CLINICAL TRIAL: NCT05966415
Title: Glycocalyx Restoration in Chronic Heart Failure: a Proof of Concept, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Endocalyx for Heart Failure
Acronym: GLYCO-HF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Rik Olde Engberink, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL81588.018.22
Record Dates: First submitted 2023-03-30; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chronic Heart Failure
Keywords: Glycocalyx; Glycosaminoglycans; Non-osmotic sodium storage; Chronic heart failure

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocalyx Pro (Experimental): Endocalyx is a food supplement that is distributed by Microvascular Health Solutions LLC in Alpine, Utah.
  Patients will receive 4 capsules Endocalyx per day, for 8 consecutive weeks. The capsules are orally administered and can be taken with water, on an empty stomach or with food.
  If possible, the patient will take 2 capsules in the morning, and 2 capsules in the afternoon. If preferred by the patient, the 4 capsules could also be taken once daily in the morning.
  Interventions: Dietary Supplement: Endocalyx Pro
- Placebo (Placebo Comparator): Placebo pills will be provided by Microvascular Health Solutions and are matched with the Endocalyx capsules. The placebo capsules contain no active pharmaceutical ingredients and contain solely widely used excipients.
  Patients will receive 4 capsules of the placebo per day for 8 consecutive weeks. The capsules are orally administered and can be taken with water, on an empty stomach or with food. If possible, the patient will take 2 capsules in the morning, and 2 capsules in the afternoon. If preferred by the patient, the 4 capsules could also be taken once daily in the morning.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Endocalyx Pro — 4 capsules once daily OR 2 capsules twice daily.
  Other Names: Endocalyx
  Arms: Endocalyx Pro
Other: placebo — 4 capsules once daily OR 2 capsules twice daily
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled study is to assess whether the food supplement Endocalyx Pro reduces sodium and water excess in patients with chronic heart failure.

The main questions it aims to answer are:

1. To assess whether the food supplement Endocalyx reduces sodium and water excess in patients with chronic heart failure.
2. To determine the contribution of different potential working mechanisms of Endocalyx in heart failure patients.
3. To evaluate whether the food supplement Endocalyx will improve patient-reported outcomes such as fluid overload symptoms and quality of life.
4. To confirm the previously demonstrated safety of Endocalyx in subjects with chronic heart failure.

Participants will be randomized to Endocalyx Pro or Placebo daily for 8 weeks, and will be followed 12 weeks.

DETAILED DESCRIPTION:
Primary Objective:

1. To assess whether the food supplement Endocalyx Pro™ (further termed Endocalyx) reduces sodium and water excess in patients with chronic heart failure.

Secondary Objectives:

1. To evaluate whether Endocalyx will improve physical limitations and patient-reported outcomes such as fluid overload symptoms and quality of life.
2. To determine the working mechanisms of Endocalyx in heart failure patients.

   1. To determine whether Endocalyx will alter tissue sodium content.
   2. To analyze whether Endocalyx reduces total body water and body weight.
   3. To assess whether Endocalyx affects office blood pressure, 24-hour blood pressure, peripheral resistance and cardiac output.
   4. To assess whether Endocalyx improves microcirculation characteristics.
   5. To evaluate whether Endocalyx reduces systemic inflammation and monocyte activation.
3. To confirm safety of Endocalyx in the heart failure population a. To compare the incidence of (serious) adverse events between Endocalyx and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Documented or suspected heart failure with reduced ejection fraction (HFrEF and HFmrEF according to ESC guidelines).
2. Signs of congestion, defined as:

   a. Elevated NT-proBNP levels: i. >450 pg/ml in subjects aged <55 years. ii. >900 pg/ml in subjects aged 55-75 years. iii. >1800 pg/ml in subjects aged >75 years. AND b. Use of diuretics, OR c. Presence of peripheral edema, OR d. Complaints of orthopnea or paroxysmal nocturnal dyspnea, OR e. A chest X-rays with sings of volume overload, OR f. Hypertension, as defined by an office blood pressure >140/90 mmHg.
3. Stable diuretic and antihypertensive treatment for the previous 3 weeks.
4. Subject, or legal representative, has voluntarily signed and dated an Informed Consent Form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.

Rationale for the inclusion criteria:

(1-3) To select the adequate subject population with appropriate disease severity for the evaluation. NT-proBNP levels are known to increase with age.(21, 22) The cutoffs of NT-proBNP levels were selected according the 2021 European Society of Cardiology Guidelines for the diagnosis and treatment of acute and chronic heart failure. (23) (4) In accordance with GCP.

Should inclusion prove difficult, we will lower required NT-proBNP levels by 25% to respectively 338, 675 and 1350 pg/ml. We will notify the METC of this decision.

Exclusion Criteria:

1. Age <18 years.
2. Estimated glomerular filtration rate (eGFR) <15 ml/min/1.73m2 measured by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
3. Systolic (<105 mmHg) or diastolic hypotension (<60 mmHg) as measured by office blood pressure measurements.
4. Severe symptoms of (orthostatic) hypotension.
5. An acute coronary syndrome, stroke, transient ischemic attack or cardiovascular surgery in the last 3 months.
6. Hospitalization for heart failure in the past 3 weeks.
7. Dialysis treatment or expected initiation of dialysis within 3 months of screening.
8. Women of child bearing potential.
9. Planned surgery in the next 8 weeks.
10. Major surgery in the previous 4 weeks.
11. Use of any other investigational drug.
12. Presence of significant comorbidities (e.g., advanced malignancy, advanced liver disease) with a life expectancy of less than 1 year.
13. A psychiatric, addictive or any disorder that compromises ability to give truly informed consent for participation in this study.
14. Known hypersensitivity to seaweed, corn, artichoke, grape, melon or to any of the excipients of Endocalyx.
15. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose galactose malabsorption.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percent change of NT-proBNP from baseline to week 8 in Endocalyx treated patients when compared with subject receiving Placebo | 8 weeks
  Our primary outcome will be the degree of volume overload as measured by the change in NT-proBNP from baseline to the study end at 8 weeks. We will compare the proportional change in NT-proBNP from baseline (as defined by the geometric mean of the screening and week 0 visit) to week 8 in a logarithmic scale using an analysis of covariance (ANCOVA). Treatment will be included in the model as fixed factor, and gender (male versus female) and baseline NT-proBNP as covariates.
  Our primary analysis will be an intention-to-treat analysis. To check the robustness of our results, we will perform a per protocol analysis. Subjects that withdraw their consent and stop the study medication will be asked to consent for a NT-proBNP measurement at the scheduled end of the study.
  NT-proBNP will be measured at screening visit, week 0 (randomization), week 4 and 8

SECONDARY OUTCOMES:
Change in 24 hour blood pressure, daytime blood pressure, nighttime blood pressure in Endocalyx treated patients when compared with subject receiving Placebo | 8 weeks
  24-hour ambulatory blood pressure (systolic blood pressure, diastolic blood pressure and mean arterial blood pressure) will be measured at screening, week 4 and week 8
Change in total body water in Endocalyx treated patients when compared with subject receiving Placebo | 8 weeks
  Total body water and body weight will be measured with a body composition monitor at week 0 (randomization visit), 4 and 8
Change in body weight (in kilograms) in Endocalyx treated patients when compared with subject receiving Placebo | 8 weeks
  Body weight will be measured at week 0 (randomization visit), 4 and 8
Change in hemodynamic parameters in Endocalyx treated patients when compared with subject receiving Placebo | 8 weeks
  Nexfin will be used to measure hemodynamic parameters (such as heart rate, cardiac output and total peripheral resistance) at week 0 (randomization visit), 4 and 8
Concentration change of Adrenomedullin in Endocalyx treated patients when compared with subject receiving Placebo | 0-8 weeks
  Adrenomedullin concentrations willl be measured in plasma. Blood will be collected at visits 0,1,2 and 3 (week 0-8)
Change/difference in ratio of classical (CD14++/CD16-), non-classical (CD14+/CD16++) and intermediate (CD14++/CD16+) monocyte subsets in Endocalyx treated patients when compared with subject receiving Placebo | 0-8 weeks
  will be isolated from peripheral blood mononuclear cells (PBMCs) collected at week 0 and 8
Difference in chemokine. scavenger receptors, and surface proteins associated with monocyte adhesion, migration and activation concentrations, in Endocalyx treated patients when compared with subject receiving Placebo | 8 weeks
  will be isolated from peripheral blood mononuclear cells (PBMCs) collected at week 0 and 8
Lipopolysaccharide-mediated cytokine secretion of monocytes in vitro in Endocalyx treated patients when compared with subjects receiving Placebo | 8 weeks
  will be isolated from peripheral blood mononuclear cells (PBMCs) collected at week 0 and 8
Difference in hospitalization rates due to heart failure in Endocalyx treated patients when compared with subjects receiving Placebo | 12 weeks
  (serious) adverse events will be asked regularly throughout the study (during each study visit, and telephone call)
Distance covered during the 6 minute walking tests in Endocalyx treated patients when compared with subjects receiving Placebo | 8 weeks
  Difference and change in meters covered during the six minute walking tests will be assessed during visit 0 (week 0) and 3 (week 8)
Change in self-reported Quality of life in Endocalyx treated patients when compared with subjects receiving Placebo | 8 weeks
  Quality of life assessment with the RAND-36 and the Dutch version of the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The MLHFQ is one of the most widely used instruments for evaluating health-related quality of life in heart failure patients internationally and has been recommended by a systematic and reliable expert-based evaluation of available heart failure-specific health-related quality of life questionnaires.
  Questionnaires will be filled in at week 0,4an 8
Difference in incidence of (serious) adverse events in Endocalyx treated patients when compared with subjects receiving Placebo | 12 weeks
  (serious) adverse events will be asked regularly throughout the study (during each study visit, and telephone call)
Pharmacokinetics of Endocalyx | 0-8 weeks
  (precursors of) glycosaminoglycans will be measured in urine and blood at set timepoints in a subset of patients who give additional informed consent at week 0,4 and 8
Skin sodium content in skin biopsies | 0-8 weeks
  In a subset of patients who give additional informed consent for skin biopsies, skin sodium content will be measured.
  Changes and differences in Endocalyx treated patients will be compared with subjects receiving Placebo.
  Skin biopsies will be taken at week 0 and 8.
monocyte and macrophage expression and density in skin biopsies | 0-8 weeks
  In a subset of patients who give additional informed consent for skin biopsies the migration of monocytes, skin macrophage density and expression will be assessed.
  Changes and differences in Endocalyx treated patients will be compared with subjects receiving Placebo.
  Skin biopsies will be taken at week 0 and 8.
Change/difference in blood pressure in Endocalyx treated patients when compared with subjects receiving Placebo | 12 weeks
  Office blood pressure (systolic and diastolic blood pressure) will be measured (standardized) during each study visit.
Difference/Change in 24-hour urine sodium and potassium excretion in Endocalyx treated patients when compared with subjects receiving Placebo | 8 weeks
  Subjects will collect 24-hour urine for the visits 1 and 3 (week 0 and 8 respectively)
Plasma aldosterone and renin change/difference in Endocalyx treated patients when compared with subjects receiving Placebo | 8 weeks
  Blood will be collected at visits 0,1,2 and 3 (week 0-8)
Differential treatment effects of Endocalyx in male and female patients | 12 weeks
  Exploratory subgroup analyses are planned to evaluate differential treatment effects of Endocalyx in male and female patients. Previous studies have demonstrated that women have lower skin sodium content than men and show less of an increase in skin sodium content after a high sodium diet.(36, 37) Also, heart failure is different in men and women. Women are more likely to have a non-ischemic ideology and hypertension as a cause of heart failure, and respond differently to treatment.(38) Considering these important gender differences in both heart failure characteristics and the suggested working mechanism of Endocalyx, it is likely that Endocalyx will have different effects in men and women.
Percent change in antihypertensive drug dosage or number prescribed | 8 weeks
  % change in antihypertensive drug dosage or number prescribed in Endocalyx treated patients when compared with subjects receiving Placebo. Medication will be reviewed during visits 0-3 and during the telephone calls
Percent change in diuretics (dosage or number prescribed) | 8 weeks
  % change in diuretics (dosage or number prescribed) prescribed in Endocalyx treated patients when compared with subjects receiving Placebo. Medication will be reviewed during visits 0-3 and during the telephone calls

CONTACTS AND LOCATIONS:
Overall Officials: Rik Olde Engberink, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided